CLINICAL TRIAL: NCT04649268
Title: The Effect of Virtual Reality and DVD Optokinetic Stimulation Exposure on Visual Induced Dizziness Symptoms in Persons With a Vestibular Disorder
Brief Title: Comparison of Optokinetic Stimulation Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC Reference: 20/LO/1244
Record Dates: First submitted 2020-11-13; First posted 2020-12-02 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2020-11

CONDITIONS: Peripheral Vestibular Disorder
Keywords: optokinetic stimulation; visually induced dizziness; vestibular; virtual reality; Oculus Quest headset

STUDY DESIGN:
Intervention Model Description: This will be a pilot study and 24 participants will be randomised into one of two rehabilitation groups incorporating OKS treatment with Optokinetic DVD (Group A) or VR headset (e.g. Oculus Quest headset) (Group B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optokinetic stimulation treatment with visual motion DVDs (Active Comparator): Customised vestibular rehabilitation programme which includes optokinetic stimulation treatment with visual motion DVDs
  Interventions: Other: Group A
- Optokinetic stimulation treatment with Virtual Reality (Experimental): Customised vestibular rehabilitation programme which includes optokinetic stimulation treatment with Virtual Reality environments delivered with headset (e.g. Oculus Quest headset)
  Interventions: Device: Group B

INTERVENTIONS:
Device: Group B — The C2 CARE C2 Physio 2019.2 has been developed for physiotherapy rehabilitation purposes including vestibular disorders. Virtual reality environments will be provided via the VR Oculus Quest headset as part of the OKS exposure incorporated within a customised VRT programme. Participants will attend 45 minute individualised supervised sessions once weekly for 8 weeks. Participants in this rehabilitation group will also have a home-based exercise programme to practise on days not attending clinic. The home-based programme will incorporate customised VRT exercises with exposure to VR environments using the VR Oculus Quest headset.
  Other Names: C2CARE Class I medical device: virtual environments; C2CARE PSY: C2 Physio 2019.2; Optokinetic stimulation treatment with Virtual Reality
  Arms: Optokinetic stimulation treatment with Virtual Reality
Other: Group A — Optokinetic stimulation treatment delivered through visual motion DVDs. Individualised 45 minute supervised sessions will occur for this group also once weekly for 8 weeks together with a home-based customised VRT programme incorporation the DVD to practise on days not attending clinic. Participants will have to use the OKS DVD for their exercises at home daily for 8 weeks as part of the prescribed home exercise programme.
  Other Names: Optokinetic stimulation treatment with visual motion DVDs
  Arms: Optokinetic stimulation treatment with visual motion DVDs

SUMMARY:
Persons with a vestibular (e.g. inner ear) disorder often report visual induced dizziness (ViD) symptom (i.e. postural and/or gait instability, dizziness, disorientation) provocation or exacerbation in environments with busy or conflicting visual motion including crowds and supermarkets. ViD is frequently associated with high disability levels, prolonged illness and poorer clinical outcome. Thus, effective treatment is a priority. Vestibular rehabilitation incorporating structured exposure to Optokinetic Stimulation (OKS) (e.g. a form of computer based intervention that involves the observation of moving visual targets to encourage visual scanning) significantly improves ViD symptoms with similar improvement noted for both 'low-tech' OKS provided via a DVD or a 'high-tech', expensive, full-field stimulus. No studies have investigated if 'lower-tech', cheaper Virtual Reality (VR) systems may be beneficial in treating ViD symptoms and whether these VR systems are more effective than an OKS DVD. The first aim of this work is to compare the effect of an OKS DVD vs "lower-tech" VR system on ViD symptoms in persons with a chronic peripheral vestibular disorder aged 18-50 years old. This study may help to identify more optimal treatment strategies in persons with a vestibular disorder.

DETAILED DESCRIPTION:
Background People with ViD report symptom (i.e. postural and/or gait instability, dizziness, disorientation) provocation or exacerbation in environments with busy or conflicting visual motion including crowds, supermarkets and scrolling computer screens. Visual dependence and impaired sensory re-weighting have been identified as main contributors to balance problems in persons with vestibular disorders and are frequently associated with high disability levels, prolonged illness, and poorer clinical outcome in adults with vestibular dysfunction including vestibular migraine.

Evidence suggests that ViD symptoms respond well to rehabilitation incorporating structured exposure to OKS. Treatment with gradual, progressive exposure to OKS in combination with static and dynamic functional balance exercises has been shown to improve visual dependency, functional balance and gait as well as symptoms provoked or exacerbated in busy visual environments, such as crowds, in persons with a vestibular disorder. It is believed that improvements in ViD following treatment with OKS is due to sensory-reweighting which is the ability of CNS to adapt its relative reliance on a specific sensory modality for purposes of orientation depending on environmental conditions, task demands and/ or pathology.

During neuroimaging studies, exposure to visual OKS, in the absence of vestibular stimulation, results in consistent activation of cortical regions involved in the control of visual motion processing and eye movement, and deactivation of parieto-insular vestibular cortices indicating a reciprocally inhibitory visual-vestibular interaction. Similarly, stimulation of multisensory vestibular cortex areas results in bilateral deactivation in visual and somatosensory cortex areas. These interactions may have a functional significance and indicate a sensor re-weighting process with greater weight given to the more reliable input thus suppressing the possible mismatch between contrasting sensory information. It is believed that the recurring exposure to conflicting visual input promotes reduced visual reliance and facilitates a more effective use of vestibule-proprioceptive cues through sensory re-weighting.

However, the exact mechanisms involved in sensory re-weighting in persons with visual induced dizziness remain poorly understood.

Finally, previous work has demonstrated that low tech OKS provided via a DVD produces the same level of improvement as a more expensive, full field stimulus. Findings for the effect of virtual reality (VR) on ViD are inconclusive. Furthermore, to date only VR provided via an immersive projection theatre, often referred to as a CAVE has been used to investigate its effect on ViD. This equipment is very expensive and available only within a specialist centre. No studies have investigated if 'lower-tech' VR such as VR headset and specifically, Oculus Quest headset, may be beneficial in treatment of ViD at a much lower cost. The use of 'lower-tech' OKS equipment is promising, more widely available to clinical practice and safe to be used at home by the patients for rehabilitation purposes. However, it is not known if one type of 'lower-tech' equipment may provide greater benefit compared to another.

Purpose of the study The proposed pilot study is a non-commercial-PhD student project. The purpose of this investigation is to compare two types of OKS based VRT for the improvement of ViD in persons with a chronic vestibular disorder.

Objectives/Aims of the study The primary objective of this study is to compare the effect of two types of optokinetic stimulation (OKS) based vestibular rehabilitation (VRT) programmes on Situational Characteristics Questionnaire (SCQ) scores in persons with a chronic vestibular disorder who experience ViD aged 18-50 years old.

The secondary objectives are to compare the pre-post treatment effect of two types of OKS based VRT on subjective dizziness, psychological state, balance confidence and objective gait, balance and ViD symptoms.

Primary Hypothesis Both types of OKS will provide significant improvement on SCQ scores, but improvement with VR will be greater.

Secondary Hypothesis VRT with VR Oculus Quest headset may provide greater treatment outcome on gait and balance control, participant's subjective symptoms, psychological state and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of a peripheral vestibular disorder;
2. chronic dizziness and/or unsteadiness;
3. 18 to 50 years old;
4. no previous rehabilitation or previous VRT programme completed with partial/no improvement;
5. willing to participate and to comply with the proposed training and testing regime; and
6. current SCQ score >0,7/4. Patient diagnosis will be based on clinical history and/or neuro-otological findings, according to published normative data and limits. Persons with Benign Paroxysmal Positional Vertigo (BPPV) will be included, in the study, due to the persistence of imbalance and dizziness after BPPV resolution. The diagnosis of migraine will be made according to the International Headache Society Criteria for Migraine as well as Neuhauser Criteria for VM.

Exclusion Criteria:

Persons with:

1. central nervous system involvement, excluding migraine. However, patients with severe migraine (> 3 migrainous headaches monthly) will be excluded.
2. fluctuating symptoms, for example, active Ménière disease;
3. acute orthopaedic disorders influencing balance control and gait;
4. a score of < 23/30 on the MoCA;
5. a score of >15/21 on the HADS for the depression component indicating significant depression symptoms;
6. inability to attend sessions;
7. diagnosis of neurological disorder;
8. currently attending or has completed a rehabilitation programme targeting balance and/or dizziness in the past year or is currently part of a clinical trial testing a medicinal product. These factors may skew both the assessment scores and treatment outcome and for this reason they are listed as exclusion criteria; and
9. lack of a good grasp of written/spoken English will be excluded. The latter due to the need to complete multiple questionnaires and the lack of funding for interpreters.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-12-28 (Estimated); Primary Completion 2021-12-28 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Situational Characteristics Questionnaire (SCQ) | Assessment of the change in this outcome will be performed at baseline (week 0) and end of treatment (week 10).
  This is the primary outcome. The Situational Characteristics Questionnaire (SCQ) -shortened version measures how frequently symptoms are provoked or exacerbated in environments with visual vestibular mismatch or intense visual motion (e.g. travelling on escalators, crowds, scrolling computer screens). Scores ≥0.7/4 indicate visual induced dizziness symptoms.

SECONDARY OUTCOMES:
Functional Gait Assessment (FGA) | Assessment of the change in this outcome will be performed at baseline (week 0) and end of treatment (week 10).
  It is a 10-item test that assesses performance on complex gait tasks (i.e. walking with head turns, stepping over an obstacle or stopping and turning). The highest score is 30 and greater outcomes are indicative of better performance. The FGA has been validated in healthy people, older adults with a history of falls and balance impairments, and people with a vestibular disorder. The minimal detectable change for the FGA is reported to be 6 points in persons with balance and vestibular disorders. Scores ≤22/30 identify fall risk and are predictable of falls in community-living older persons within 6 months.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | Assessment of the change in this outcome will be performed at baseline (week 0) and end of treatment (week 10).
  Cambridge Neuropsychological Test Automated Battery (CANTAB) is a semi-automated computer program that utilizes a touch screen technology and press pad, to assess neurocognitive function. The CANTAB core cognition battery is a validated cognitive assessment system for assessing multiple components of cognitive function, including attention, visual memory, spatial memory, executive function and reaction time.
  Each subject will be comfortably seated at approximate distance of 0.5m away from the screen pad monitor and will be asked to complete the CANTAB tests after instructions have been provided. The tests that will be included are Rapid Visual Information Processing (RVP), Paired Associates Learning (PAL), Spatial Working Memory (SWM), Reaction Time (RTI), Delayed Matching to Sample (DMS), Motor Screening Task (MOT), Spatial Span (SSP) and Multitasking Test (MTT). The test order will be different for each participant.
Rod and Disc Test | Assessment of the change in this outcome will be performed at baseline (week 0) and end of treatment (week 10).
  Visual dependence is measured using the Rod and Disk Test on a laptop computer. Participants will be seated in front of a computer in a darkened room with their head held against a viewing cone that blocks extraneous visual orientation cues. The diameter of the cone at the participants' eyes will be 15cm with a depth of field of 30 cm, subtending a viewing angle of 39 degrees. The visual stimulus consists of a luminous white 6cm rod on a black background. The rod rotated 360 degrees in either direction about its midpoint in the central 11 degrees of the visual filed. Outside of this central zone, the viewing screen is filled with a collage of 220 off-white dots, each 8mm (1.5 degrees of visual field) in diameter, randomly distributed on a black background. Participants control the orientation of the rod with a roller mouse. They are instructed to align the rod to their perceived vertical (the subjective visual vertical) under three conditions.
LEGSys™ and Balansens (Biosensics, MA, USA) | Assessment of the change in this outcome will be performed at baseline (week 0) and end of treatment (week 10).
  LEGSys™and Balansens (Biosensics, MA, USA) which will be used to assess gait and balance respectively, are a validated wearable technology that uses five inertial sensors (triaxial accelerometer and gyroscope) attached to both shins above ankles, thighs above knees, and lower back close to sacrum.
  Balance will be measured in four trials of 15 seconds, (1) with eyes open on a stable surface with no visual target specified, (2) with eyes closed on a stable surface, (3) with eyes closed on an incline surface and (4) with eyes closed on a foam surface. Gait assessment will be conducted as participants will walk a distance with a minimum of 25 steps under four conditions: (1) habitual over ground normal walk (preferred speed), (2) fast over ground, (3) habitual over ground normal walk with horizontal head turns and (4) habitual over ground normal walk with vertical head turns.
Montreal Cognitive Assessment (MoCA) Tool | Assessment of the change in this outcome will be performed at baseline (week 0) and end of treatment (week 10).
  The Montreal Cognitive Assessment (MoCA) Tool is a rapid screening tool for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive function, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. It has been recommended that a cut-off scores of 23/30 be used to identify multi-domain cognitive impairment. This is the first test that will be completed. Persons with scores <23/30 will not be included in the study and will be referred back to the clinical team for further assessment and onward referral as required.
Hospital Anxiety and Depression Scale (HADS) | Assessment of the change in this outcome will be performed at baseline (week 0) and end of treatment (week 10).
  The HADS, a 14-item scale which assesses non-somatic anxiety (HAD-A) and depression (HAD-D) symptoms, will also be completed. Scores range from 0-21 for each subscale with a score ≥8 proposed for the identification of caseness, for both depression and anxiety.
Vertigo Symptom Scale (VSS) | Assessment of the change in this outcome will be performed at baseline (week 0) and end of treatment (week 10).
  The VSS is used to assess the frequency and severity of common vestibular (VSS-V; e.g. vertigo, imbalance) and autonomic/somatic (VSS-A; e.g. heart pounding, heavy feeling in the arms or legs) symptoms. Normalised scores range from 0-4, with higher scores indicating a higher (i.e. worse) level of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

REFERENCES:
- [Result] Pavlou M, Lingeswaran A, Davies RA, Gresty MA, Bronstein AM. Simulator based rehabilitation in refractory dizziness. J Neurol. 2004 Aug;251(8):983-95. doi: 10.1007/s00415-004-0476-2. PMID 15316804
- [Result] Bisdorff A, Von Brevern M, Lempert T, Newman-Toker DE. Classification of vestibular symptoms: towards an international classification of vestibular disorders. J Vestib Res. 2009;19(1-2):1-13. doi: 10.3233/VES-2009-0343. No abstract available. PMID 19893191
- [Result] Indovina I, Riccelli R, Chiarella G, Petrolo C, Augimeri A, Giofre L, Lacquaniti F, Staab JP, Passamonti L. Role of the Insula and Vestibular System in Patients with Chronic Subjective Dizziness: An fMRI Study Using Sound-Evoked Vestibular Stimulation. Front Behav Neurosci. 2015 Dec 9;9:334. doi: 10.3389/fnbeh.2015.00334. eCollection 2015. PMID 26696853
- [Result] Lempert T. Vestibular migraine. Semin Neurol. 2013 Jul;33(3):212-8. doi: 10.1055/s-0033-1354596. Epub 2013 Sep 21. PMID 24057824
- [Result] Pavlou M, Bronstein AM, Davies RA. Randomized trial of supervised versus unsupervised optokinetic exercise in persons with peripheral vestibular disorders. Neurorehabil Neural Repair. 2013 Mar-Apr;27(3):208-18. doi: 10.1177/1545968312461715. Epub 2012 Oct 16. PMID 23077146
- [Result] Pavlou M, Kanegaonkar RG, Swapp D, Bamiou DE, Slater M, Luxon LM. The effect of virtual reality on visual vertigo symptoms in patients with peripheral vestibular dysfunction: a pilot study. J Vestib Res. 2012;22(5-6):273-81. doi: 10.3233/VES-120462. PMID 23302708
- [Result] Cawthorne TE. The physiological basis for head exercises. J Chart Soc Physiother. 1944; 30:106-107.
- [Result] Morozetti PG, Gananca CF, Chiari BM. Comparison of different protocols for vestibular rehabilitation in patients with peripheral vestibular disorders. J Soc Bras Fonoaudiol. 2011 Mar;23(1):44-50. doi: 10.1590/s2179-64912011000100011. English, Portuguese. PMID 21552732
- [Result] Whitney SL, Wrisley DM, Brown KE, Furman JM. Physical therapy for migraine-related vestibulopathy and vestibular dysfunction with history of migraine. Laryngoscope. 2000 Sep;110(9):1528-34. doi: 10.1097/00005537-200009000-00022. PMID 10983955
- [Result] Dieterich M, Bense S, Stephan T, Yousry TA, Brandt T. fMRI signal increases and decreases in cortical areas during small-field optokinetic stimulation and central fixation. Exp Brain Res. 2003 Jan;148(1):117-27. doi: 10.1007/s00221-002-1267-6. Epub 2002 Nov 13. PMID 12478402
- [Result] Kleinschmidt A, Thilo KV, Buchel C, Gresty MA, Bronstein AM, Frackowiak RS. Neural correlates of visual-motion perception as object- or self-motion. Neuroimage. 2002 Aug;16(4):873-82. doi: 10.1006/nimg.2002.1181. PMID 12202076
- [Result] Brandt T, Bartenstein P, Janek A, Dieterich M. Reciprocal inhibitory visual-vestibular interaction. Visual motion stimulation deactivates the parieto-insular vestibular cortex. Brain. 1998 Sep;121 ( Pt 9):1749-58. doi: 10.1093/brain/121.9.1749. PMID 9762962
- [Result] Shumway-Cook A, Horak FB. Rehabilitation strategies for patients with vestibular deficits. Neurol Clin. 1990 May;8(2):441-57. PMID 2193221
- [Result] Van Ombergen A, Heine L, Jillings S, Roberts RE, Jeurissen B, Van Rompaey V, Mucci V, Vanhecke S, Sijbers J, Vanhevel F, Sunaert S, Bahri MA, Parizel PM, Van de Heyning PH, Laureys S, Wuyts FL. Altered functional brain connectivity in patients with visually induced dizziness. Neuroimage Clin. 2017 Feb 28;14:538-545. doi: 10.1016/j.nicl.2017.02.020. eCollection 2017. PMID 28331800
- [Result] 15. D.S.C. Cruz-Neira & T. DeFanti, Surround-screen projection-based virtual reality: Design and implementation of the CAVE, in: Proceedings of SIGGRAPH, 1993; 135-142.
- [Result] Carson N, Leach L, Murphy KJ. A re-examination of Montreal Cognitive Assessment (MoCA) cutoff scores. Int J Geriatr Psychiatry. 2018 Feb;33(2):379-388. doi: 10.1002/gps.4756. Epub 2017 Jul 21. PMID 28731508
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Result] Davies RA, Luxon LM. Dizziness following head injury: a neuro-otological study. J Neurol. 1995 Mar;242(4):222-30. doi: 10.1007/BF00919595. PMID 7798121
- [Result] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Result] Lempert T, Olesen J, Furman J, Waterston J, Seemungal B, Carey J, Bisdorff A, Versino M, Evers S, Newman-Toker D. Vestibular migraine: diagnostic criteria. J Vestib Res. 2012;22(4):167-72. doi: 10.3233/VES-2012-0453. PMID 23142830
- [Result] Neuhauser H, Leopold M, von Brevern M, Arnold G, Lempert T. The interrelations of migraine, vertigo, and migrainous vertigo. Neurology. 2001 Feb 27;56(4):436-41. doi: 10.1212/wnl.56.4.436. PMID 11222783
- [Result] Pavlou M, Quinn C, Murray K, Spyridakou C, Faldon M, Bronstein AM. The effect of repeated visual motion stimuli on visual dependence and postural control in normal subjects. Gait Posture. 2011 Jan;33(1):113-8. doi: 10.1016/j.gaitpost.2010.10.085. Epub 2010 Dec 8. PMID 21144753
- [Result] Dichgans J, Held R, Young LR, Brandt T. Moving visual scenes influence the apparent direction of gravity. Science. 1972 Dec 15;178(4066):1217-9. doi: 10.1126/science.178.4066.1217. PMID 4637810
- [Result] Cousins S, Cutfield NJ, Kaski D, Palla A, Seemungal BM, Golding JF, Staab JP, Bronstein AM. Visual dependency and dizziness after vestibular neuritis. PLoS One. 2014 Sep 18;9(9):e105426. doi: 10.1371/journal.pone.0105426. eCollection 2014. PMID 25233234
- [Result] Najafi B, Horn D, Marclay S, Crews RT, Wu S, Wrobel JS. Assessing postural control and postural control strategy in diabetes patients using innovative and wearable technology. J Diabetes Sci Technol. 2010 Jul 1;4(4):780-91. doi: 10.1177/193229681000400403. PMID 20663438
- [Result] Najafi B, Helbostad JL, Moe-Nilssen R, Zijlstra W, Aminian K. Does walking strategy in older people change as a function of walking distance? Gait Posture. 2009 Feb;29(2):261-6. doi: 10.1016/j.gaitpost.2008.09.002. Epub 2008 Oct 25. PMID 18952435
- [Result] Aminian K, Najafi B, Bula C, Leyvraz PF, Robert P. Spatio-temporal parameters of gait measured by an ambulatory system using miniature gyroscopes. J Biomech. 2002 May;35(5):689-99. doi: 10.1016/s0021-9290(02)00008-8. PMID 11955509
- [Result] Muchna A, Najafi B, Wendel CS, Schwenk M, Armstrong DG, Mohler J. Foot Problems in Older Adults Associations with Incident Falls, Frailty Syndrome, and Sensor-Derived Gait, Balance, and Physical Activity Measures. J Am Podiatr Med Assoc. 2018 Mar;108(2):126-139. doi: 10.7547/15-186. Epub 2017 Aug 30. PMID 28853612
- [Result] Mohler MJ, Wendel CS, Taylor-Piliae RE, Toosizadeh N, Najafi B. Motor Performance and Physical Activity as Predictors of Prospective Falls in Community-Dwelling Older Adults by Frailty Level: Application of Wearable Technology. Gerontology. 2016;62(6):654-664. doi: 10.1159/000445889. Epub 2016 Apr 30. PMID 27160666
- [Result] Najafi B, Lee-Eng J, Wrobel JS, Goebel R. Estimation of Center of Mass Trajectory using Wearable Sensors during Golf Swing. J Sports Sci Med. 2015 May 8;14(2):354-63. eCollection 2015 Jun. PMID 25983585
- [Result] Thiede R, Toosizadeh N, Mills JL, Zaky M, Mohler J, Najafi B. Gait and balance assessments as early indicators of frailty in patients with known peripheral artery disease. Clin Biomech (Bristol). 2016 Feb;32:1-7. doi: 10.1016/j.clinbiomech.2015.12.002. Epub 2015 Dec 22. PMID 26775227
- [Result] Wrisley DM, Marchetti GF, Kuharsky DK, Whitney SL. Reliability, internal consistency, and validity of data obtained with the functional gait assessment. Phys Ther. 2004 Oct;84(10):906-18. PMID 15449976
- [Result] Marchetti GF, Lin CC, Alghadir A, Whitney SL. Responsiveness and minimal detectable change of the dynamic gait index and functional gait index in persons with balance and vestibular disorders. J Neurol Phys Ther. 2014 Apr;38(2):119-24. doi: 10.1097/NPT.0000000000000015. PMID 24637931
- [Result] Wrisley DM, Kumar NA. Functional gait assessment: concurrent, discriminative, and predictive validity in community-dwelling older adults. Phys Ther. 2010 May;90(5):761-73. doi: 10.2522/ptj.20090069. Epub 2010 Apr 1. PMID 20360052
- [Result] Cambridge-Cognition-Limited. CANTABeclipse™: Test Administration Guide Manual. 3rd ed. Cambridge 2015.
- [Result] Egerhazi A, Berecz R, Bartok E, Degrell I. Automated Neuropsychological Test Battery (CANTAB) in mild cognitive impairment and in Alzheimer's disease. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Apr 13;31(3):746-51. doi: 10.1016/j.pnpbp.2007.01.011. Epub 2007 Jan 16. PMID 17289240
- [Result] Fowler KS, Saling MM, Conway EL, Semple JM, Louis WJ. Paired associate performance in the early detection of DAT. J Int Neuropsychol Soc. 2002 Jan;8(1):58-71. PMID 11843075
- [Result] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Result] Yardley L, Masson E, Verschuur C, Haacke N, Luxon L. Symptoms, anxiety and handicap in dizzy patients: development of the vertigo symptom scale. J Psychosom Res. 1992 Dec;36(8):731-41. doi: 10.1016/0022-3999(92)90131-k. PMID 1432863
- [Result] Guerraz M, Yardley L, Bertholon P, Pollak L, Rudge P, Gresty MA, Bronstein AM. Visual vertigo: symptom assessment, spatial orientation and postural control. Brain. 2001 Aug;124(Pt 8):1646-56. doi: 10.1093/brain/124.8.1646. PMID 11459755
- [Result] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Result] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. In. Vol 4: J Pharmaceutical Statistics 2005; (4): 287-291.
- [Result] Micarelli A, Viziano A, Micarelli B, Augimeri I, Alessandrini M. Vestibular rehabilitation in older adults with and without mild cognitive impairment: Effects of virtual reality using a head-mounted display. Arch Gerontol Geriatr. 2019 Jul-Aug;83:246-256. doi: 10.1016/j.archger.2019.05.008. Epub 2019 May 10. PMID 31102927
- [Result] Oculus Quest Review: Facebook's VR Savior Mostly Keeps its Promises. UploadVR 2019-05-22. Retrieved 2019-06-02.
- [Result] Pavlou M, Davies RA, Bronstein AM. The assessment of increased sensitivity to visual stimuli in patients with chronic dizziness. J Vestib Res. 2006;16(4-5):223-31. PMID 17538212
- [Result] Viziano A, Micarelli A, Augimeri I, Micarelli D, Alessandrini M. Long-term effects of vestibular rehabilitation and head-mounted gaming task procedure in unilateral vestibular hypofunction: a 12-month follow-up of a randomized controlled trial. Clin Rehabil. 2019 Jan;33(1):24-33. doi: 10.1177/0269215518788598. Epub 2018 Jul 16. PMID 30012022
- [Result] Park JH, Jeon HJ, Lim EC, Koo JW, Lee HJ, Kim HJ, Lee JS, Song CG, Hong SK. Feasibility of Eye Tracking Assisted Vestibular Rehabilitation Strategy Using Immersive Virtual Reality. Clin Exp Otorhinolaryngol. 2019 Nov;12(4):376-384. doi: 10.21053/ceo.2018.01592. Epub 2019 May 9. PMID 31066247